CLINICAL TRIAL: NCT07090499
Title: A Phase 1 Open-label Study to Investigate PF-08046876 in Adult Participants With Advanced Solid Tumors.
Brief Title: A Study to Learn About the Study Medicine Called PF-08046876 in People With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5951001; 2025-521729-33-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Advanced/Metastatic Solid Tumors; Bladder Cancer; Urothelial Carcinoma; Advanced Non-Small Cell Lung Cancer; Carcinoma, Non Small Cell Lung; Carcinoma, Squamous Cell of Head and Neck; Head and Neck Cancer; Esophageal Cancer; Gastroesophageal Junction Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Esophageal Adenocarcinoma; Pancreatic Adenocarcinoma; Pancreatic Cancer
Keywords: B6C; integrin beta 6; ADC; antibody drug conjugate; bladder cancer; urothelial carcinoma; non-small cell lung cancer; NSCLC; head and neck cancer; HNSCC; SCCHN; esophageal cancer; EC; esophageal squamous cell carcinoma; gastroesophageal junction adenocarcinoma; pancreatic cancer; PDAC; pancreatic adenocarcinoma; esophageal adenocarcinoma; lung adenocarcinoma; lung squamous cell carcinoma; integrin alpha-v beta-6 receptor; ITGB6
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus; Pancreatic Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Escalation (Experimental): Different groups of participants will receive different doses and/or schedules of the study drug
  Interventions: Drug: PF-08046876
- Part 2 Dose Optimization (Experimental): Participants will be randomized to 2 dosing regimens deemed to be safe in Part 1
  Interventions: Drug: PF-08046876
- Part 2 Dose Expansion (Experimental): Participants in tumor-specific groups will receive 1 dosing regimen deemed to be safe in Part 1
  Interventions: Drug: PF-08046876

INTERVENTIONS:
Drug: PF-08046876 — Intravenous administration

SUMMARY:
The purpose of the study is to explore the safety and effects of the study drug (PF-08046876) in people diagnosed with advanced cancer of the bladder, lung, head and neck, esophagus, or pancreas. PF-08046876 is an investigational anticancer therapy called an 'antibody drug conjugate' or 'ADC'. ADCs are anticancer drugs designed to stick to cancer cells and kill them.

The study drug will be given to participants through a needle in a vein (intravenous infusion). This study includes multiple parts. In the first part of the study, there will be different groups of people receiving different doses of the study drug. The study may also test different schedules.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Advanced cancer of the bladder, lung, head and neck, esophagus, or pancreas
* Measurable disease
* ECOG Performance status 0-1
* Part 1: progression or relapse following standard treatments
* Part 2: maximum of 2 prior lines of systemic therapy in the advanced setting
* Resolution of acute effects of prior anticancer therapy to baseline or Grade 1
* Consent to submit required pre-treatment tumor tissue as medically feasible

Exclusion criteria:

* Received prior treatment with an antibody drug conjugate with a camptothecin-class payload (e.g. sacituzumab govitecan, trastuzumab deruxtecan )
* Active anorexia, nausea or vomiting, and/or signs of intestinal obstruction meeting protocol exclusion
* Pulmonary disease meeting protocol exclusion
* Other unacceptable abnormalities as defined by protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-07-08 (Estimated); Study Completion 2029-07-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) estimated during the Adverse Events (AE) evaluation | Start of treatment up to 30 days after last dose or start of new anticancer therapy (whichever occurs first)
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy dose modifications.
Part 1: Number of Participants With Dose-limiting Toxicities (DLTs): Monotherapy | Baseline to end of DLT evaluation period
  Occurrence of DLTs as defined by the protocol
Part 1: Recommended Monotherapy Dose for Expansion | Baseline to 30 days post last study drug administration
  RDE will be based on cumulative safety, preliminary antitumor activity and pharmacokinetics findings
Part 2: Recommended Phase 2 Dose | Baseline to 30 days post last study drug administration
  RP2D will be determined based on the cumulative safety, preliminary anti tumor activity and Pharmacokinetics findings.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until the date of the first documentation of disease progression, death, or start of new anticancer therapy (approximately 2 years)
  ORR defined as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Duration of Response (DOR) | From the date of the first objective response to the date of disease progression or death (approximately 2 years)
  DOR as defined per RECIST 1.1.
Progression Free Survival (PFS) | From Baseline to date of first disease progression or death (approximately 2 Years)
  PFS as defined per RECIST 1.1.
Overall Survival (OS) | From baseline to up to 3 years
  OS defined as the time until death due to any cause.
Pharmacokinetics (PK): Maximum Observed Serum Concentration (Cmax) | Baseline to approximately 30 days after last dose of study drug
  Evaluate the single and multiple dose PK of PF-08048676.
PK: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Baseline to approximately 30 days after last dose of study drug
  Evaluate the single and multiple dose PK of PF-08048676.
PK: Area Under the Curve (AUC) from Time Zero to Last Quantifiable Concentration (AUClast) | Baseline to approximately 30 days after last dose of study drug
  Evaluate the single and multiple dose PK of PF-08048676.
Incidence of Anti-Drug Antibody (ADA) | Baseline to approximately 30 days after last dose of study drug
  To evaluate the immunogenicity of PF-08046876.
Incidence of Neutralizing Antibodies (NAb) | Baseline to approximately 30 days after last dose of study drug
  To evaluate the immunogenicity of PF-08046876.
Percent change of immune cells within tumors based on multiplex immunofluorescence | Baseline through 4-7 weeks after first dose of study drug
  This measure will assess changes in the presence or activation of immune cells in the tumor microenvironment using RNA and/or Immunohistochemistry (IHC) assays.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (11):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center - Conroe, Conroe, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center - West Houston, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center - League City, League City, Texas
  - NEXT Oncology, San Antonio, Texas
  - The University of Texas, MD Anderson Cancer Center - Sugar Land, Sugar Land, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5951001